CLINICAL TRIAL: NCT01899456
Title: A Randomized Safety and Efficacy Study Investigating the Effects of Catheter-based Renal Denervation in Patients After Renal Transplantation
Brief Title: Impact of Sympathetic Renal Denervation- a Study in Patients After Renal Transplantation
Acronym: ISAR-denerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Simon Schneider, Simon Schneider, MD; 1.Medizinische Klinik und Poliklinik, Klinikum rechts der Isar, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5548/12
Record Dates: First submitted 2013-07-10; First posted 2013-07-15 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension; Chronic Kidney Disease; Renal Transplantation; Sympathetic Activity
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical therapy (No Intervention): Best medical therapy using guideline recommended drugs in each disease state.
- Catheter-based renal denervation (Experimental): Renal denervation will be performed in the native renal arteries of patients after renal transplantation. Access side is the contralateral femoral artery.
  Interventions: Device: Catheter-based renal denervation

INTERVENTIONS:
Device: Catheter-based renal denervation
  Other Names: Renal denervation with Symplicity Catheter Medtronic/Ardian
  Arms: Catheter-based renal denervation

SUMMARY:
The study is aiming to document the safety and effectiveness of renal denervation in patients after renal transplantation with hypertension. Catheter-based renal denervation will be performed using CE marked, percutaneous Symplicity catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patient after renal transplantation (> 6 month) without resection of native kidneys
* systolic blood pressure >=150 mmHg
* on 3 or more antihypertensive medications
* Individual is 18 years of age
* Individual agrees to have all procedures performed, and is competent and willing to provide written, informed consent to participate in the registry.

Exclusion Criteria:

* secondary causes and a white coat hypertension
* renal artery abnormalities
* eGFR < 30mL/min (MDRD)
* angina
* severe Aortic valve stenosis
* Individual is pregnant, nursing or planning to be pregnant
* other

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-07; Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of renal denervation in patients after renal transplantation | Baseline to 6 months
  Effect on blood pressure including office, ABPM, and home-based measurements. Number of adverse events. Changes of antihypertensive medications. Effects on renal function assessed with glomerular filtration rate. Renovascular safety (renal artery stenosis) assessed by duplex ultrasound.

SECONDARY OUTCOMES:
Effect of renal denervation in patients after renal transplantation on different organ systems. | Baseline to 6 month
  Effects on sympathetic activity assessed by heart rate variability and post extrasystolic potentiation. Glucose metabolism and insulin resistance (fasting and during oGTT). Hospitalization rates (eg. hypertensive emergencies, heart failure, etc).

CONTACTS AND LOCATIONS:
Overall Officials: Simon Schneider, MD, Principal Investigator — 1. Medizinische Klinik und Poliklinik, Klinikum rechts der Isar, Technische Unversität München
Locations (1):
- 1. Medizinische Klinik und Poliklinik, Klinikum rechts der Isar, Technische Universität München, Munich, Germany

REFERENCES:
- [Result] Schneider S, Promny D, Sinnecker D, Byrne RA, Muller A, Dommasch M, Wildenauer A, Schmidt G, Heemann U, Laugwitz KL, Baumann M. Impact of sympathetic renal denervation: a randomized study in patients after renal transplantation (ISAR-denerve). Nephrol Dial Transplant. 2015 Nov;30(11):1928-36. doi: 10.1093/ndt/gfv311. Epub 2015 Sep 1. PMID 26333545